CLINICAL TRIAL: NCT00415883
Title: An Open-Label, Randomized, Single Dose, Two Period, Crossover Study to Determine the Relative Bioavailability of Valsartan 160 mg Japanese Formulation and Valsartan 160 mg Global Formulation in Healthy Adult Volunteers
Brief Title: To Compare the Blood Level of Marketed Japanese Valsartan Tablet Formulation vs Global Valsartan Tablet Formulation in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CVNP489A2106
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Healthy
Keywords: Relative bioavailability, formulation, Japanese, valsartan, healthy subjects
MeSH Terms: interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Valsartan

SUMMARY:
The purpose of this study is to assess how the body changes the blood level of single dose of valsartan 160 mg tablet Japanese formulation and valsartan 160 mg tablet global formulation under fasting condition in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male or female subjects age 18 to 45 years of age (inclusive)
* In good health
* Female subjects either surgically sterilized at least 6 months prior to study participation or post-menopausal (no regular menstrual bleeding for at least 2 years)
* Body mass index within the range of 18.5 to 28 kg/m2 and weigh at least 45 kg

Exclusion Criteria:

* Smokers
* Use prescription drugs within 4 weeks prior dosing, or over-the-counter medication (vitamins, herbal supplements, dietary supplements, potassium supplements) within 2 weeks prior to dosing. Paracetamol is acceptable
* Participation in any clinical investigation within 4 weeks prior to dosing
* Donation or loss of 400 mL or more of blood within 8 weeks prior to first dosing
* Significant illness within 2 weeks prior to dosing.
* History of clinically significant cardiac abnormalities, fainting, low blood pressure upon standing, irregular heartbeats.
* History of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or untreated).
* History of clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis).
* Known hypersensitivity or severe reaction to valsartan or similar drugs
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize the subject in case of participation in the study.
* History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
* History of drug or alcohol abuse within the 6 months prior to dosing

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2006-07

PRIMARY OUTCOMES:
Relative bioavailability of valsartan 160 mg Japanese formulation and valsartan 160 mg global formulation under fasting conditions in healthy adult volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, Mumbai, India